CLINICAL TRIAL: NCT04657757
Title: Investigation of Bacterial Adhesion and Bactericide Effect ex Vivo on Different Implant Restoration Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-00248; sp20Zeller
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Dental Diseases
Keywords: intraoral biofilm formation; parodontitis; tooth implant; periimplant diseases
MeSH Terms: conditions — Stomatognathic Diseases; Dry Socket

STUDY DESIGN:
Masking Description: The test persons are numbered so that the laboratory technician who performs the analysis of the platelets cannot be assigned a name. Blinding with regard to the materials is not possible, as the color differences of the alloys allow for a classification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoral apparatus (Experimental): intraoral apparatus in which two platelets of each of the 8 materials (Esteticor Lumina PF; Esteticor Lumina PF - after Lactic acid storage; Pagalinor 2; Esteticor Economic; Pekkton ivory - untreated; Pekkton ivory - rough; Oralloy; Machined Titan Zirconia (TiZr) alloy) are to be examined. Examination is a crystal violet OD595 staining (10 minutes). The color absorbed by the bacteria is then dissolved with a 30% acetic acid and measured spectrophotometrically at 595 nm. The plaque formed on the material surface is removed immediately after removal from the oral cavity and analyzed by determination of Colony Forming Unit (CFU) number.
  Interventions: Other: Intraoral apparatus

INTERVENTIONS:
Other: Intraoral apparatus — Eight platelets with different material composition and surface properties are fastened in a holder (carrier rondell) with 15 mm diameter and inserted into the braces. Braces are to be worn for 28 hours in the oral cavity except for meals and oral hygiene procedures. Platelets then are removed and analyzed. After a first course the braces are to be cleaned in chlorhexidine solution in an ultrasonic bath; followed by a second identical course (Braces to be worn for 28 hours in the oral cavity except for meals and oral hygiene procedures).

SUMMARY:
Investigation of bacterial adhesion and bactericide effect ex vivo on different implant restoration materials

DETAILED DESCRIPTION:
The aim of this study is to investigate bacterial attachment and bactericidal effects of different materials used for the transmucosal part of implants. Using a brace, the intraoral biofilm formation in healthy subjects will be measured after 28 hours (24 hours intraorally, 4 hours rest). For this purpose 2 sterile platelets of each of the 8 differently processed materials (16 platelets in total) are inserted into the braces.

The main target parameter is the quantification of the biofilm by crystal violet staining. For this purpose the samples are analyzed by spectrophotometry at a wavelength of 595 nm (OD595).

As secondary target parameter possible bactericidal effects of the materials, which are analyzed by Colony forming units (CFU) determination, are used.

ELIGIBILITY:
Inclusion Criteria:

* No systemic antibiotic therapy during the last 3 months
* Good oral hygiene and compliance (plaque index (PI) <20%, bleeding index (BI) <20%)
* No signs of periodontitis or other inflammatory changes in surrounding tissues
* Non-smokers

Exclusion Criteria:

* Disease that requires antibiotics
* Pressure points caused by the braces, which cannot be eliminated by adjusting
* Other unforeseen complications that can be associated with braces

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
quantification of biofilm | 2x 24hours in a period of about 10 days
  quantification of the biofilm by crystal violet staining. For this purpose the samples are analyzed by spectrophotometry at a wavelength of 595 nm (OD595).

SECONDARY OUTCOMES:
number of CFU | 2x 24hours in a period of about 10 days
  Possible bactericidal effects of the materials, which are analyzed by CFU determination, serve as secondary target parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Zitzmann, MD PhD, Principal Investigator — University Center for Dentistry Basel UZB
Locations (1):
- University Center for Dentistry Basel UZB, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No